CLINICAL TRIAL: NCT00918164
Title: A Randomized, Open-Label, Single Dose, Crossover Study To Evaluate The Relative Bioavailability Of PF-04457845 Tablet To Solution Formulation And To Assess Food Effect In Healthy Subjects
Brief Title: Evaluation Of The Relative Bioavailability Of PF-04457845 Tablet To Solution Formulation And Food Effect In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B0541005
Record Dates: First submitted 2009-05-05; First posted 2009-06-11 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy adult volunteers (Experimental): Standard Phase 1 normal healthy adult volunteers, age range 21-55 years and of either sex
  Interventions: Drug: PF-04457845

INTERVENTIONS:
Drug: PF-04457845 — Single dose, 8 mg as oral tablet and solution formulation

SUMMARY:
The purpose of this study is to estimate the bioavailability of PF-04457845 tablets relative to solution and evaluate the effect of food (fasted vs. high fat meal) on the pharmacokinetics of an oral tablet formulation of PF-04457845

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or healthy female subjects of non-child bearing potential. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests);
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs);
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial;
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures;
* Willing and able to consume a non-vegetarian high-fat meal.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
* History of febrile illness within 5 days prior to the first dose;
* Any condition possibly affecting drug absorption (eg, gastrectomy);
* A positive urine drug screen;
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening;
* Treatment with an investigational drug within 30 days or 5 half-lives (or determined by the local requirement, whichever is longer) preceding the first dose of trial medication;
* 12-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility;
* Pregnant or nursing females and females of child-bearing potential;
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication;
* Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of trial medication. Other exceptions may be granted by a qualified member of Pfizer study management;
* Unwillingness to refrain from consumption of grapefruit/pomelo or grapefruit/pomelocontaining products from 7 days prior to the first dose of study medication until the completion of the follow-up visit.
* Blood donation of approximately 1 unit (~500 mL) within 56 days prior to dosing;
* Unwillingness or inability to comply with the Lifestyle guidelines;
* Subject is the Investigator or sub-Investigator, research assistant, pharmacist, study coordinator, other staff, or a relative of study personnel directly involved with the conduct of the study;
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics | up to 96 hours post dose

SECONDARY OUTCOMES:
Safety and toleration including adverse events, vital signs measurements, 12-lead ECGs, Physical examination findings, Blood and urine safety tests. | pre-dose to follow up

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0541005&StudyName=Evaluation%20Of%20%20The%20Relative%20Bioavailability%20Of%20PF-04457845%20Tablet%20To%20Solution%20Formulation%20And%20Food%20Effect%20In%20Healthy%20Subjects